CLINICAL TRIAL: NCT00921076
Title: Gait Analysis of Patients Undergoing Total Ankle Arthroplasty, Ankle Arthrodesis, Tibiotalocalcaneal or Pantalar Fusion.
Brief Title: Gait Analysis of Ankle Arthroplasty and Arthrodesis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMH 02-035
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2009-07

CONDITIONS: Ankle Arthritis
MeSH Terms: interventions — Gait Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ankle Arthoplasty (Active Comparator): Patients will undergo a Total Ankle Replacement procedure
  Interventions: Behavioral: Gait Analysis
- Ankle fusion (Active Comparator): Patients will undergo an Ankle Arthrodesis procedure
  Interventions: Behavioral: Gait Analysis

INTERVENTIONS:
Behavioral: Gait Analysis — A computerized motion analysis system to observe the effect of ankle arthroplasty versus ankle arthrodesis on the kinematic behaviour of the foot and ankle during gait.

SUMMARY:
Surgical options for managing hindfoot arthritis include: joint fusion, total ankle joint replacement or osteotomies (realignment) of bones. Fusion of arthritic hindfoot joints has been the accepted method of managing hindfoot arthritis for over a century. Recently, total ankle replacement has evolved as a treatment option for patients with end stage ankle arthritis. A comparison of gait for patients before and after hindfoot fusion or total ankle replacement will give further information about the outcome of this treatment. The principal aim of this project is to assess the effect of total ankle replacement or hindfoot fusion on gait. We are also interested in the outcome of the surgery and its effect on your symptoms (eg. pain and mobility). The results of this study will aid researchers in assessing this new treatment modality. Your involvement in this study is critical for the researchers to further analyze this new form of treatment and your time and involvement is appreciated.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic Ankle Arthritis
2. Skeletal maturity
3. Able to give informed consent

Exclusion Criteria:

1. Avascular Necrosis of Talus
2. Obesity (BMI >30)
3. Prior Ankle fusion or arthroplasty
4. Active or prior infection within 12 months
5. Medical condition precluding major surgery
6. Severe ipsilateral mid or hind foot deformity
7. Severe osteoporotic or osteopenic bone
8. Neuromuscular impairment
9. Age less than 40 years old
10. Cognitive or psychiatric impairment prohibiting accurate follow-up
11. Pregnancy
12. Workers compensation board patients

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2002-06; Primary Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure will be micro motion, consisting of component migration and rotation relative to the talus and distal tibia. This will be measured utilizing RSA with bi-planar stereo X-rays taken at several intervals: before weight bearing is | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Timothy R. Daniels, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada